CLINICAL TRIAL: NCT01321892
Title: Ex Vivo Multimodal Imaging of Upper Aerodigestive Epithelium
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: William Marsh Rice University (Other)
Responsible Party: Sponsor
Other Study IDs: GCO # 09-0945
Record Dates: First submitted 2011-03-21; First posted 2011-03-24 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Squamous Cell Carcinoma of the Oral Cavity; Oropharynx; Larynx; Hypopharynx
Keywords: HRME; High-resolution microendoscope; Optical imaging technology; Non-invasive fluorescence and reflectance imaging; Upper aerodigestive tract; Cancer surgery; Squamous cell carcinoma; Oral cavity; Oropharynx; Larynx; Hypopharynx; Squamous cell carcinoma of the oral cavity, oropharynx, larynx, and/or hypopharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Laryngeal Diseases; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Retained specimens are punch biopsy specimens from the primary tumor resection.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Squamous cell carcinoma: Patients included in this study will be receiving surgical treatment for their biopsy-proven squamous cell carcinoma.

SUMMARY:
The purpose of this research study is to collect information on whether images made using investigational microscopes can improve researchers' ability to evaluate and distinguish between normal and abnormal areas in tissue samples surgically removed from patients with squamous cell carcinoma. The microscopes being used in this study are considered investigational because they have not been approved by the United States Food and Drug Administration (FDA) for finding abnormal or pre-cancerous areas.

DETAILED DESCRIPTION:
The overall objective of this exploratory study is to evaluate whether noninvasive fluorescence and reflectance imaging of the upper aerodigestive tract can help clinicians more accurately determine intraoperative margins during ablative cancer surgery. This is an ex vivo study designed to evaluate the feasibility of using prototype optical imaging technology to enhance the discrimination between areas of noncancerous "normal" and cancerous mucosa. The results of this laboratory study will be used to further refine and develop this technology for in vivo application.

Primary Aim:

(1) To collect data to develop imaging algorithms to distinguish between normal and cancerous upper aerodigestive mucosa.

Secondary Aims:

1. To compare the combination of wide-field fluorescence/reflectance and high resolution fluorescence microscopy images of upper aerodigestive epithelium to histopathologic analysis of biopsied tissue.
2. To compare the ability of sequential wide-field/fluorescence microscopy imaging to discriminate between normal and cancerous oral cavity mucosa with that of white-light images obtained after staining with toluidine blue.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with biopsy-proven squamous cell carcinoma of the oral cavity, oropharynx, larynx, and/or hypopharynx.
* Must be receiving surgical treatment for their cancer.

Exclusion Criteria:

• Presence of medical or psychiatric condition affecting ability to give voluntary, informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with new head and neck cancer, who reside in the tri-state area.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2009-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Accuracy and Interrater Reliability of HRME Image Interpretation | baseline
  We will ask blinded raters to classify the HRME images as either benign (normal) or dysplastic/cancerous (abnormal)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sikora, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Blair EA, Callender DL. Head and neck cancer. The problem. Clin Plast Surg. 1994 Jan;21(1):1-7. PMID 8112003
- [Background] Silverman S Jr, Sugerman PB. Oral premalignancies and squamous cell carcinoma. Clin Dermatol. 2000 Sep-Oct;18(5):563-8. doi: 10.1016/s0738-081x(00)00146-2. No abstract available. PMID 11134851
- [Background] Schwarz RA, Gao W, Daye D, Williams MD, Richards-Kortum R, Gillenwater AM. Autofluorescence and diffuse reflectance spectroscopy of oral epithelial tissue using a depth-sensitive fiber-optic probe. Appl Opt. 2008 Feb 20;47(6):825-34. doi: 10.1364/ao.47.000825. PMID 18288232
- [Background] Ramanujam N, Mitchell MF, Mahadevan A, Warren S, Thomsen S, Silva E, Richards-Kortum R. In vivo diagnosis of cervical intraepithelial neoplasia using 337-nm-excited laser-induced fluorescence. Proc Natl Acad Sci U S A. 1994 Oct 11;91(21):10193-7. doi: 10.1073/pnas.91.21.10193. PMID 7937860
- [Background] Gillenwater A, Jacob R, Richards-Kortum R. Fluorescence spectroscopy: a technique with potential to improve the early detection of aerodigestive tract neoplasia. Head Neck. 1998 Sep;20(6):556-62. doi: 10.1002/(sici)1097-0347(199809)20:63.0.co;2-o. PMID 9702544
- [Background] Pavlova I, Weber CR, Schwarz RA, Williams MD, Gillenwater AM, Richards-Kortum R. Fluorescence spectroscopy of oral tissue: Monte Carlo modeling with site-specific tissue properties. J Biomed Opt. 2009 Jan-Feb;14(1):014009. doi: 10.1117/1.3065544. PMID 19256697
- [Background] Epstein JB, Zhang L, Poh C, Nakamura H, Berean K, Rosin M. Increased allelic loss in toluidine blue-positive oral premalignant lesions. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2003 Jan;95(1):45-50. doi: 10.1067/moe.2003.97. PMID 12539026
- [Background] Epstein JB, Sciubba J, Silverman S Jr, Sroussi HY. Utility of toluidine blue in oral premalignant lesions and squamous cell carcinoma: continuing research and implications for clinical practice. Head Neck. 2007 Oct;29(10):948-58. doi: 10.1002/hed.20637. PMID 17764090
- [Background] Martin IC, Kerawala CJ, Reed M. The application of toluidine blue as a diagnostic adjunct in the detection of epithelial dysplasia. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1998 Apr;85(4):444-6. doi: 10.1016/s1079-2104(98)90071-3. PMID 9574954
- [Background] Kerawala CJ, Beale V, Reed M, Martin IC. The role of vital tissue staining in the marginal control of oral squamous cell carcinoma. Int J Oral Maxillofac Surg. 2000 Feb;29(1):32-5. PMID 10691141
- [Background] Genden EM, Desai S, Sung CK. Transoral robotic surgery for the management of head and neck cancer: a preliminary experience. Head Neck. 2009 Mar;31(3):283-9. doi: 10.1002/hed.20972. PMID 18972413
- [Background] McNeil BJ, Weichselbaum R, Pauker SG. Speech and survival: tradeoffs between quality and quantity of life in laryngeal cancer. N Engl J Med. 1981 Oct 22;305(17):982-7. doi: 10.1056/NEJM198110223051704. PMID 7278922
- [Background] Collier T, Lacy A, Richards-Kortum R, Malpica A, Follen M. Near real-time confocal microscopy of amelanotic tissue: detection of dysplasia in ex vivo cervical tissue. Acad Radiol. 2002 May;9(5):504-12. doi: 10.1016/s1076-6332(03)80326-4. PMID 12458875
- [Background] Muldoon TJ, Pierce MC, Nida DL, Williams MD, Gillenwater A, Richards-Kortum R. Subcellular-resolution molecular imaging within living tissue by fiber microendoscopy. Opt Express. 2007 Dec 10;15(25):16413-23. doi: 10.1364/oe.15.016413. PMID 19550931
- [Background] Feuer EJ, Kessler LG. Test statistic and sample size for a two-sample McNemar test. Biometrics. 1989 Jun;45(2):629-36. PMID 2765642
- [Background] Rosenberg D, Cretin S. Use of meta-analysis to evaluate tolonium chloride in oral cancer screening. Oral Surg Oral Med Oral Pathol. 1989 May;67(5):621-7. doi: 10.1016/0030-4220(89)90286-7. PMID 2654801